CLINICAL TRIAL: NCT06298786
Title: Validation and Evaluation of the Mastication Function in Adults: The Functional Six-minute Mastication Test (F-6MMT).
Acronym: F-6MMT
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Universitària del Bages (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: F6MMT_JPA
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Mastication Disorder; Fatigue; Temporomandibular Disorder; Orofacial Pain; Chewing Problem
MeSH Terms: conditions — Fatigue; Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Subjects with TMD Screener score < 3
  Interventions: Diagnostic Test: Functional 6-minute mastication test
- TMD subjects: Subjects with TMD screener score ≥ 3
  Interventions: Diagnostic Test: Functional 6-minute mastication test

INTERVENTIONS:
Diagnostic Test: Functional 6-minute mastication test — All participants will be evaluated in 3 different phases. First, they will respond to the online TMD screener questionnaire. Then, they will be presentally evaluated using the DC/TMD and finally they will undergo the functional 6-minute mastication test.
  Other Names: TMD-Screener; Diagnostic criteria for temporomandibular disorders (DC/TMD)

SUMMARY:
Temporomandibular Disorders (TMD) encompass various conditions that affect the temporomandibular joint and associated tissues, often causing or being associated with other symptoms such as jaw pain, myofascial pain, neck pain, and headaches. TMDs are classified according to the DC/TMD instrument in which the joint and pain axes are evaluated. However, there is no evaluation of mandibular function, and TMDs can result in a decrease in jaw strength and resistance. This leads to an increase in the chewing fatigue. Reliable and time-effective diagnostic methods for evaluating masticatory function are crucial in the clinical setting because of the high prevalence of TMD. Chewing efficiency is essential for food preparation and nutrient absorption, and muscle fatigue is a common problem affecting chewing ability. Despite this, there is a lack of validated tests to evaluate chewing fatigue in patients with TMD, which makes its consideration unnoticed in clinical practice.

The modified six-minute functional chewing test (F-6MMT) was proposed as a tool to evaluate chewing ability and fatigue in patients with TMD. This test is an adaptation of a previously designed test in which subjects with mitochondrial pathology were evaluated; however, the subjects were not instructed to perform functional chewing during the test. In this version, modifications are added so that the test is as functional as possible, allowing chewing to be evaluated in a standardized way, and cut-off points established between healthy subjects and subjects with TMD in terms of chewing capacity in general and fatigue in particular. This study will follow standardized reporting guidelines and recruit participants from diverse clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Women and men of legal age
* With or without TMDs symptoms and
* With or without self-reported jaw fatigue when eating

Exclusion Criteria:

* Subjects treated with any type of treatment requiring infiltration of the mandibular region
* Participants undergoing dental interventions in the last 3 months
* Individuals missing two or more teeth in the same quadrant.
* Inability to understand or speak catalan, spanish or english.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents from the Central region of Catalonia and Vallès Occidental, and patients from the University Clinics of the UIC and UVic-UCC, Campus Manresa.
Sampling Method: Probability Sample
Enrollment: 514 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Immediately before the procedure, immediately after the procedure, and five minutes after the procedure
  Score fatigue on a Numerical Rating Scale (0-10). 0 means no fatigue and 10 the highest fatigue possible.
Self-reported Pain | Immediately before the procedure, immediately after the procedure, and five minutes after the procedure
  Score pain on a Numerical Rating Scale (0-10). 0 means no pain and 10 the highest pain possible
Sensitivity and Specificity | through study completion, an average of 1 year
  Ability to identificate cases vs controls
Feasibity | through study completion, an average of 1 year
  Intra and inter examinator feasibility
Replicability | Through study completion, an average of 1 year
  Consistency and precision of the test

SECONDARY OUTCOMES:
Pain-related TMD diagnosis | Before the procedure
  All subjects will be classified into the following categories according to the diagnostic criteria for temporomandibular disorders: i) positive TMD (TMD-P), ii) arthralgia (TMD-A), iii) local myalgia (TMD-LM), iv) myofascial pain (TMD-MP), v) headache attributed to TMDs (TMD-HA) or vi) negative TMD (TMD-N)
Self-reported daily fatigue | Baseline
  Dichotomous answers (YES/NO) from the question: "Do you feel tension, heaviness, tiredness, or fatigue of the jaw muscles in any of the daily activities such as chewing, eating, swallowing, smiling, kissing, gesturing, smiling, singing or yawning?"
Pain pressure threshold (PPT) | Immediately before the procedure, immediately after the procedure, and five minutes after the procedure
  For measuring PPT a digital algometer (Baoshinshan), with a precision ± 0,2% and a metallic extremity of one cm2 will be used at masseter, anterior temporalis, and forearm of both sides. Scores of the PPT will be measured as Kg/cm^2
Taste of the gum | Immediately after the procedure
  Score taste on a Numerical Rating Scale (0-10). 0 means not tasty, and 10 absolutely tasty.
Preferred side when chewing during the F-6MMT | Immediately after the procedure
  Score how easy was to chew the gum for each side. Numerical Rating Scale (0-10). 0 means preferred left side, 5 means balanced, and 10 preferred right side.
Kinesiofobia related to TMD | Before the procedure
  Questionnaire TSK-TMD. Score from 12 to 48 points
Health status | Before the procedure
  Patient Health Questionnaire-4 (PHQ-4). Score from 0 to 12.
Comorbidities | Before the procedure
  Central Sensitization Inventory. Score from 0 to 125 and a checklist

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Clinica Universitaria UManresa - UViv-UCC, Campus Manresa, Manresa, Barcelona
  - Universitat de Manresa, Manresa, Barcelona
  - Universitat Internacional de Catalunya, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scrivani SJ, Keith DA, Kaban LB. Temporomandibular disorders. N Engl J Med. 2008 Dec 18;359(25):2693-705. doi: 10.1056/NEJMra0802472. No abstract available. PMID 19092154
- [Background] Sheikholeslam A, Moller E, Lous I. Pain, tenderness and strength of human mandibular elevators. Scand J Dent Res. 1980 Feb;88(1):60-6. doi: 10.1111/j.1600-0722.1980.tb00721.x. PMID 6929087
- [Background] Svensson P, Arendt-Nielsen L, Houe L. Muscle pain modulates mastication: an experimental study in humans. J Orofac Pain. 1998 Winter;12(1):7-16. PMID 9656894
- [Background] Wozniak K, Lipski M, Lichota D, Szyszka-Sommerfeld L. Muscle fatigue in the temporal and masseter muscles in patients with temporomandibular dysfunction. Biomed Res Int. 2015;2015:269734. doi: 10.1155/2015/269734. Epub 2015 Mar 26. PMID 25883949
- [Background] van der Bilt A, Engelen L, Pereira LJ, van der Glas HW, Abbink JH. Oral physiology and mastication. Physiol Behav. 2006 Aug 30;89(1):22-7. doi: 10.1016/j.physbeh.2006.01.025. Epub 2006 Mar 29. PMID 16564557
- [Background] Gisel EG. Chewing cycles in 2- to 8-year-old normal children: a developmental profile. Am J Occup Ther. 1988 Jan;42(1):40-6. doi: 10.5014/ajot.42.1.40. PMID 3354628
- [Background] Koutris M, Lobbezoo F, Naeije M, Wang K, Svensson P, Arendt-Nielsen L, Farina D. Effects of intense chewing exercises on the masticatory sensory-motor system. J Dent Res. 2009 Jul;88(7):658-62. doi: 10.1177/0022034509338573. PMID 19641154
- [Background] Farella M, Bakke M, Michelotti A, Martina R. Effects of prolonged gum chewing on pain and fatigue in human jaw muscles. Eur J Oral Sci. 2001 Apr;109(2):81-5. doi: 10.1034/j.1600-0722.2001.00991.x. PMID 11347660
- [Background] Castroflorio T, Falla D, Tartaglia GM, Sforza C, Deregibus A. Myoelectric manifestations of jaw elevator muscle fatigue and recovery in healthy and TMD subjects. J Oral Rehabil. 2012 Sep;39(9):648-58. doi: 10.1111/j.1365-2842.2012.02309.x. Epub 2012 Apr 10. PMID 22490056
- [Background] Le Reverend BJ, Edelson LR, Loret C. Anatomical, functional, physiological and behavioural aspects of the development of mastication in early childhood. Br J Nutr. 2014 Feb;111(3):403-14. doi: 10.1017/S0007114513002699. Epub 2013 Sep 24. PMID 24063732
- [Background] van den Engel-Hoek L, Knuijt S, van Gerven MH, Lagarde ML, Groothuis JT, de Groot IJ, Janssen MC. The 6-min mastication test: a unique test to assess endurance of continuous chewing, normal values, reliability, reproducibility and usability in patients with mitochondrial disease. J Oral Rehabil. 2017 Mar;44(3):155-162. doi: 10.1111/joor.12481. Epub 2017 Jan 30. PMID 28054362
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Bossuyt PM, Cohen JF, Gatsonis CA, Korevaar DA; STARD group. STARD 2015: updated reporting guidelines for all diagnostic accuracy studies. Ann Transl Med. 2016 Feb;4(4):85. doi: 10.3978/j.issn.2305-5839.2016.02.06. No abstract available. PMID 27004232
- [Background] Gonzalez YM, Schiffman E, Gordon SM, Seago B, Truelove EL, Slade G, Ohrbach R. Development of a brief and effective temporomandibular disorder pain screening questionnaire: reliability and validity. J Am Dent Assoc. 2011 Oct;142(10):1183-91. doi: 10.14219/jada.archive.2011.0088. PMID 21965492
- [Background] González Y, Rivera Y, Espinosa I. Adaptación transcultural de los criterios diagnósticos para la investigación de los trastornos temporomandibulares (CDI/TTM). Rev Fac Odontol Univ Antioq. 2013;25:11-25
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Visscher CM, Lobbezoo F, Naeije M. Comparison of algometry and palpation in the recognition of temporomandibular disorder pain complaints. J Orofac Pain. 2004 Summer;18(3):214-9. PMID 15509000
- [Background] Calixtre LB, Oliveira AB, Alburquerque-Sendin F, Armijo-Olivo S. What is the minimal important difference of pain intensity, mandibular function, and headache impact in patients with temporomandibular disorders? Clinical significance analysis of a randomized controlled trial. Musculoskelet Sci Pract. 2020 Apr;46:102108. doi: 10.1016/j.msksp.2020.102108. Epub 2020 Jan 11. PMID 31999615
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Herr K, Spratt KF, Garand L, Li L. Evaluation of the Iowa pain thermometer and other selected pain intensity scales in younger and older adult cohorts using controlled clinical pain: a preliminary study. Pain Med. 2007 Oct-Nov;8(7):585-600. doi: 10.1111/j.1526-4637.2007.00316.x. PMID 17883743
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520